CLINICAL TRIAL: NCT07208396
Title: UPPER CERVICAL MOBILIZATION VERSUS INTEGRATED NEUROMUSCULAR INHIBITION TECHNIQUE IN PATIENTS WITH LEVATOR SCAPULAE SYNDROME
Acronym: LSS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Ebrahem Sadek, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005854
Record Dates: First submitted 2025-09-24; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Levator Scapulae Syndrome
Keywords: trigger points

STUDY DESIGN:
Intervention Model Description: The Integrated Neuromuscular Inhibition Technique (INIT) is an approach that combines three interventions: Ischemic Compression, Strain Counter Strain, and Muscle Energy Technique. INIT aims to stretch the fascia and muscle structures and increase muscle flexibility, prevent and eliminate taut bands/trigger points and adhesions on the fascia, eliminate complaints of pain and headaches, reduce stiffness, and improve functional abilities .
  Cervical mobilization is the common approach used by physical therapists to treat mechanical neck pain using manual therapy, it aims to enhance tissue extensibility, increase range of motion (ROM), mobilize soft tissue or joints, and reduce pain. Cervical mobilization has been shown to be an effective treatment for mechanical neck pain .
  conventional physical therapy will be in the form of: (superficial heat using hot pack for 10 minutes , Isometric Neck Exercises and Dynamic Neck
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UPPER CERVICAL MOBILIZATION (Experimental): All patients in group A will receive Grades I and II mobilizations and conventional physical therapy program in the form of :( hot pack, Dynamic and Isometric Neck Exercises) for four weeks.
  Interventions: Other: Upper cervical mobilization
- Integrated neuromuscular inhibition technique (Experimental): Group B will receive integrated neuromuscular inhibition Technique and conventional physical therapy program as in group A in the form of :( hot pack, Dynamic and Isometric Neck Exercises) for four weeks.
  Interventions: Other: Integrated neuromuscular inhibition technique
- conventional treatment (Active Comparator): Participants in group C will receive conventional physical therapy only in the form of: (superficial heat using hot pack for 10 minutes, Dynamic Neck Exercises and Isometric Neck Exercises) for four weeks
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Upper cervical mobilization — All patients in group A will receive Grades I and II mobilizations in the first two sessions to reduce pain. In subsequent sessions, patients will receive Grades III and IV mobilizations; typically will be utilized to stretch the joint capsule and passive tissues, which provide stability to the joint, thereby increasing ROM. Maitland usually performs treatment techniques in an oscillatory manner. These oscillations can be performed with different amplitudes in different positions in the range of movement.
  The mobilizations will be delivered in the prone position. The duration of mobilization will be 30-s bouts given for three sets. The therapist places a hand dorsally at the level of the vertebral arch of C1 with the metacarpophalangeal and radial border of the index finger. The other hand will be placed posteriorly under the occiput, with the shoulder positioned anteriorly on the patient's forehead. The mobilization force will be directed dorsally from the shoulder until the therapist
  Arms: UPPER CERVICAL MOBILIZATION
Other: Integrated neuromuscular inhibition technique — An integrated approach to myofascial trigger point release is achieved by combining several manual therapy techniques under the name INIT (Integrated Neuromuscular Inhibition Technique). The technique combines MET and SCS with ischemic compression in one coordinated technique .
  First, intermittent compression(IC) was initiated by using the thumb and index finger to apply a pincer grip to the TrP in the middle of the UT.
  Second, the strain counter strain (SCS) began by applying pressure to the trigger point . The participants' heads were passively flexed laterally to the affected side. and then asked the patient about pain.
  Third, the MET begins with one of the investigator's hands stabilizing the affected shoulder and the other on the head side. The participant was asked to move the stabilized shoulder and head in the direction of the other. This contraction lasted 7 seconds and had a maximum voluntary contraction of 20%. After that, the muscle was lengthened for 30 seconds
  Arms: Integrated neuromuscular inhibition technique
Other: Conventional treatment — 1. Hot packs Hot pack will be applied at the beginning of the treatment session for all patients participated in the study. The participants will be in prone lying position. The neck and upper thoracic region will be exposed. The hot pack then will be applied for 10 minutes on cervical and upper thoracic region.
  2. Dynamic neck exercise: Dynamic neck exercises include lifting head up with the chin tucked in from supine lying for neck flexion, lifting head backwards in prone lying for neck extension lifting head sideways from pillow in side lying position for neck side flexion which will be also repeated for the other side.
  3. Isometric Neck Exercises The exercises will be performed in sitting position, by holding the theraband directly forwards for neck flexion, backwards for neck extension and obliquely towards right and left and by crossing over the band for neck side flexion and rotation. All these will be done for all patients participated in the study for about 5-10 repetition
  Arms: conventional treatment

SUMMARY:
the study will be conducted to answer the following research question: is there a difference between the effect of upper cervical mobilization and integrated neuromuscular inhibition technique of levator scapulae muscle in patients with levator scapulae syndrome?

DETAILED DESCRIPTION:
Neck pain might be usually provoked by TrPs in the upper trapezius and levator scapulae muscles The differentiation in levator scapulae MTrPs prevalence between the right and left sides may also indicate potential asymmetries in muscle use or stress, which could be relevant for diagnosis and treatment strategies.

Integrated treatment approach (INIT) for neck pain provides greater pain relief, reduces disability, improves functional ability, and improves quality of life than other treatments Cervical Spine Mobilization (CSM) by oscillatory movements and traction to the cervical segments helps to break adhesion and stretch the hypo-mobile shortened structures.

There is a gap in the available literature about the comparative effect of upper cervical mobilization and integrated neuromuscular inhibition technique (INIT) of levator scapulae muscle on neck pain, neck disability, range of motion, and cervical proprioception in levator scapulae syndrome.

60 Participants recruited from both genders will be assigned randomly into 3 equal groups Group A : will receive upper cervical mobilization plus conventional treatment .

Group B : will receive integrated neuromuscular technique, It is a technique which combines three methods (Ischemic compression- muscle energy technique- strain counter strain) plus conventional treatment .

Group C : will receive conventional physical therapy only in the form of: (superficial heat using hot pack for 10 minutes ,Isometric Neck Exercises and Dynamic Neck) .

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a primary complaint of chronic neck pain (assessed by VAS) for more than 3 months.
2. Subjects with pain provocation and reduced mobility at the upper cervical segment (assessed by passive accessory intervertebral movements (PAIVMs) and reduced mobility at cervical spine (assessed by CROM) will be included in the study.
3. Participants will be recruited from both genders with age ranged from 18 to 45 years old, and BMI from 18 to 30kg/m2

Exclusion Criteria:

* 1) Previous spine surgery 2) Pregnant and breast feeding women 3) Diabetic patients 4) Hypertensive patients 5) Neck pain associated with cervical radiculopathy 6) Whiplash injuries 7) Cervical spine fracture 8) Vertebrobasilar insufficiency. 9) Red flags suggesting of cancer, infection, vascular insufficiency

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
pain pressure threshold of trigger points | up to 4 weeks
  The Pressure Pain Threshold (PPT) is defined as the point at which a non-painful pressure stimulus turns into a painful pressure sensation. Pressure algometry (PA) is a method described to objectify this PPT. This technique is a well-known and well-validated method to induce acute experimental pain. Different studies have been published about using this tool to evaluate pain in different locations of the body and showed high levels of reliability.
Measurement of Neck Functional Disability Level using the Arabic Version of Neck Disability Index | up to 4 weeks
  The patient will be relaxed and asked to complete the NDI before treatment and after treatment, which consists of 10 items. Each item is scored from zero (no disability) to five (total disability), with the maximum possible total score being 50. For each item, the subject asked to choose one answer that best defined his/her neck functional disability level. Scores for each item tallied and the total score will be recorded. Mean duration of the test: 3 to 7.8 minutes. Vernon and Mior presented the following interpretation

SECONDARY OUTCOMES:
Measurement of cervical proprioception | up to 4 weeks
  Most assessment techniques currently available evaluate the integrity and function of efferent pathways or the final outcome of skeletal muscle activation or a combination of both Joint position sense is one dimension of proprioception, classically assessed by the ability to accurately reproduce preselected target positions or a specific joint angle . The test usually involves some type of position matching procedure, in which a target joint position is presented and the subject must match that position. The absolute difference between the target and the matching joint positions is often used as a measure of position sense accuracy in terms of the repositioning error.
Range of motion assessment of cervical spine | up to 4 weeks
  Cervical active range of motion (AROM) in flexion and extension, right/left side bending and right/left rotation will be measured for each subject.